CLINICAL TRIAL: NCT06011356
Title: Smart Watch Insights for Prevention of Exacerbations and Enhance Rehabilitation - Movement Study
Acronym: SWIPER-MOVES
Status: Active, not recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 22HH7499
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Cardiovascular Diseases; Non-Alcoholic Fatty Liver Disease; Respiratory Disease; Diabetes
Keywords: Digital health; Smart wearable; Population health; Digital biomarkers
MeSH Terms: conditions — Cardiovascular Diseases; Non-alcoholic Fatty Liver Disease; Respiration Disorders; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Smartwatch — Activity tracker (step count, calories burned), measures heart rate, heart variability and other physiological variables.

SUMMARY:
Aims of the study:

1. To deliver a scalable wellbeing programme to the local population of Imperial College Healthcare NHS Trust, focusing on movement.
2. To describe the natural history of long-term conditions using digital data from a smartwatch.
3. To identify digital information that is routinely collected by a smart watch that can be used to predict outcomes in patients with long term conditions.
4. To identify factors that determine whether participants engage with and improve in a movement programme.

Adult patients who are registered to the Imperial NHS Care Information Exchange (CIE), an NHS patient-facing electronic health record, are eligible to participate in the study. Participants will receive a smart watch for self-monitoring of their movement and wellbeing and be asked to wear the device as much as possible. They will be asked to download a smartphone application called Connected Life, which displays movement and information on heart rate, breathing and oxygen levels to both the participant and the research team (digital data). Participants will receive secure login details for the Connected Life application from the research team, to ensure data privacy. The research team will look at participants' health records, and attempt to identify associations between the digital data and clinical information. This will allow the research team to identify digital data that predicts the onset and natural history of long term conditions, which may potentially allow for earlier diagnosis for future patients. The primary outcome of the study is the identification of trends in movement based on step-count data recorded by the smartwatch.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years
* Registered with the patient-facing electronic health record (Care Information Exchange)

Exclusion Criteria:

* Unwilling or unable to provide informed consent
* Arm or wrist injury or condition prohibiting the safe use of a smartwatch
* Any visual impairment preventing the use of the smartwatch or smartphone application.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will recruit study participants from patients registered to the Imperial College Healthcare NHS Trust Care Information Exchange (CIE), a patient-facing electronic health record. Patients on CIE have already provided consent to be approached for NHS research.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Step count | 24 months
  Change and trends in step count

SECONDARY OUTCOMES:
Quality of life (EQ-5D-5L) | 24 months
  Change in quality of life as measured by the EQ-5D-5L questionnaire
Patient Activation Measure (PAM) | 24 months
  Change in patient engagement and confidence over own health, as measured by the Patient Activation Measure

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas S Peters, MD, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom (+44), United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided